CLINICAL TRIAL: NCT00209612
Title: Phase I/II Study of Biweekly Administration Regimen of Paclitaxel Combined With CPT-11 in Patients With Second Line Chemotherapy of Inoperable or Recurrent Gastric Cancer(GC).
Brief Title: Phase I/II Study of Paclitaxel Plus CPT-11 in Pts. With 2nd Line Chemotherapy of Inoperable or Recurrent GC.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: due to strong side effect
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Collaborators: Hokkaido University Hospital (Other)
Responsible Party: Yoshito Komatsu / A vice-director, Associate Prof., Hokkaido University Hospital Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0402; PacIri
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Paclitaxel+Irinotecan
  Interventions: Drug: Taxol; Drug: Campt, Topotesin

INTERVENTIONS:
Drug: Taxol — Day1,15 X mg/m2, IV (in the vein)
  Other Names: Paclitaxel
Drug: Campt, Topotesin — Day1,15 Y mg/m2, IV (in the vein)
  Other Names: irinotecan

SUMMARY:
A phase I/II study is conducted to determine the maximum-tolerated dose (MTD), dose-limiting toxicity (DLT), and efficacy of a combination chemotherapy using CPT-11 and Paclitaxel in pre-treated patients with metastatic gastric cancer. The usefulness of the this regimen is evaluated by response rate, median survival time, and progression free survival.

DETAILED DESCRIPTION:
Patients with pre-treated measurable metastatic gastric cancer were included in this trial. Patients received this combination chemotherapy repeated every 28 days until progression disease. Starting dose (dose level 1) were CPT-11 80 mg/m2 on day 1 and 15, Paclitaxel 60 mg/m2 on day 1 and 15. DLT was defined as follows (according to NCI-CTC version 2.0); Grade 4 neutropenia, thrombocytopenia(≥25000), Grade 3 neutropenia accompanied fever (>38℃) , and Grade 3 non-hematological toxicity (except for nausea, vomit, appetite loss , general fatigue, alopecia). Maximal Tolerated Dose (MTD) is determined when the incidence of critical toxicity exceeds 50% at a certain dose level. Response rate will be calculated according to RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or recurrent gastric cancer with prior treatment for advanced disease.
* Patients who have received 1cycle cancer therapy (radiotherapy, chemotherapy or chemoradiotherapy) given > 4 weeks prior to the beginning of study therapy
* At least one measurable lesion according to the RECIST criteria. Minimum indicator lesion size: > 10 mm measured by spiral CT or >20mm measured by conventional techniques(Except for Phase I setting).
* Patients aged between 20 and 75 years, inclusive, at the time of acquisition of informed consent
* Patients with performance status(ECOG) 0 to 2
* Abnormal hematologic values (WBC ≥ 3.5 x 109/L, Hemoglobin ≥ 9.0g/dl, platelet count ≥ 100 x 109/L)
* Serum cleatinine ≤ 1.5mg/dl
* Serum bilirubin ≤ 1.5mg/dl. ALT, AST ≤ 2.0 x upper normal limit (or ≤ 3 x upper normal limit in the case of liver metastases)
* Normal ECG
* Life expectancy ≥ 3 months
* Patients who have given written informed consent to participate in this study

Exclusion Criteria:

* Patients with active multiple cancers; or even if the multiple cancers are metachronous, have a disease-free period of less than 5 years (but excluding cancer in situ and skin cancer) (Except for Phase I setting)
* Serious, uncontrolled, concurrent infection(s) or illness(es)
* Patients with no serious concurrent complications (such as heart disease, Intestinal pneumonia)
* Patients with Liver cirrhosis
* Patients with fresh hemorrhage from the gastrointestinal tract
* Patients with poorly controlled diabetes or are treated by continuous use of insulin
* Patients with concurrent psychiatric disease or psychotic symptoms, and judged to have difficulties participating in the study
* Patients with retention of body fluid(pleural effusion, ascites, pericardial effusion) necessitating treatment
* Patients with diarrhea (watery stool)
* Patients with infection, intestinal palsy or intestinal occlusion
* Patients with brain metastasis
* Patients with Gilbert syndrome
* Patients who have experienced serious drug allergy in the past
* Patients who are pregnant and lactating or hope to become pregnant during the study period
* Patients with prior Taxan (Paclitaxel, Docetaxel) or CPT-11 treatment
* Patients with neuropathy ≥ grade 2
* Others, patients judged by the investigator or subinvestigator to be inappropriate as subject

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-04; Primary Completion 2008-11 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Determine the DLT(Dose Limiting Toxicity) and MTD(Maximum Tolerated Dose) in Phase I setting. Determine the clinical response rate with Recommended dose in Phase II setting. | 1-year

SECONDARY OUTCOMES:
Determine the clinical response rate of patients in Phase I setting. | 1-year
Determine the MST(Median Survival Time) and PFS(Progression Free Survival) in Phase II setting. | 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Asaka, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- ・ Hokkaido University Hospital (Hokkaido University Graduate School of Medicine / School of Medicine), Sapporo, Hokkaido, Japan